CLINICAL TRIAL: NCT04079257
Title: The Pharmacokinetics and Pharmacodynamics of Eculizumab in Patients With Paroxysmal Nocturnal Hemoglobinuria
Acronym: PREPARE
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: PREPARE
Record Dates: First submitted 2019-07-11; First posted 2019-09-06 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria; Eculizumab; PK-PD
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with paroxysmal nocturnal hemoglobinuria: Patients are already treated with eculizumab. The only intervention is the collection of extra blood samples to measure peak concentrations of eculizumab
  Interventions: Other: Blood collection for measurement of eculizumab peak concentrations

INTERVENTIONS:
Other: Blood collection for measurement of eculizumab peak concentrations — collection of blood
  Other Names: blood collection

SUMMARY:
Because of the inter and intra individual variability in pharmacokinetics and pharmacodynamics of eculizumab in PNH patients, a tailored treatment approach for the individual is probably preferable. The starting point of a robust tailored dosing approach for eculizumab is the development of a population pharmacokinetic-pharmacodynamic model. In this cross-sectional observational pharmacokinetic and pharmacodynamic study, trough and peak concentrations of eculizumab are measured to describe the pharmacokinetics and complement activation markers to describe the pharmacodynamics.

DETAILED DESCRIPTION:
Paroxysmal nocturnal hemoglobinuria (PNH) is a rare hematological disorder which is characterized by hemolytic anemia, cytopenias and thrombosis. PNH is caused by clonal expansion of hematopoietic stem cells with an acquired somatic mutation in the X-linked phosphatidylinositol glycan class A gene (4). This gene encodes a protein required for synthesis of glycosylphosphatidylinositol (GPI) anchors. As a result of the mutation, affected stem cells are deficient in GPI anchored proteins. Clonal expansion leads to the production of hematological cells lacking the expression of GPI anchored complement regulatory proteins CD55 and CD59.

This leads to chronic complement-mediated hemolysis of the GPI-deficient erythrocytes. Eculizumab is a humanized chimeric monoclonal anti-C5 inhibitor which is approved for the treatment of PNH and was the first licensed drug targeting the complement system. By binding to C5, eculizumab prevents the activation of C5 into C5a and C5b and subsequent the formation of the terminal complement complex C5b-9. Eculizumab is currently administered in a flat fixed dose for every patient. However, because of the inter and intra individual variability in pharmacokinetics and pharmacodynamics of eculizumab in PNH patients, a tailored treatment approach for the individual is probably preferable. We have recently shown, by means of pharmacokinetic modelling and simulation, based on the drug approval data, that eculizumab dosing in PNH patients can be successfully tailored by means of Therapeutic Drug Monitoring.

This approach when implemented in practice will result in overall less pharmacokinetic variability, less under-treatment and an average dose reduction of 11%. It should be noted that the yearly eculizumab drug costs are about 400.000 euro per patient. Considering the fact that in the Netherlands alone approximately 60 patients with PNH are yearly treated with this drug, this indicates that development of a model-informed precision dosing tool based on the actual pharmacokinetics and pharmacodynamics of eculizumab has the potential to decrease treatment costs with 2.640.000 euro on a yearly basis. The starting point of a robust tailored dosing approach for eculizumab is the development of a population pharmacokinetic-pharmacodynamic model. The majority of the pharmacokinetic and pharmacodynamic data in PNH patients are derived from controlled clinical studies and may not be representative for general PNH patient population. Therefore, it is pivotal to collect more pharmacokinetic and pharmacodynamic data in PNH patients in the actual clinical setting.

This study is a cross-sectional observational pharmacokinetic study in which we collect trough and peak concentrations of eculizumab to describe the pharmacokinetics and complement activation markers to describe the pharmacodynamics. With this data, a pharmacokinetic-pharmacodynamic model will be developed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PNH
* Treated with eculizumab
* Willing to give informed consent

Exclusion Criteria:

* Not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PNH patients treated with eculizumab
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Clearance | 9 months
  Peak and trough concentrations will be measured in order to determine clearance
Volume of distribution | 9 months
  Peak and trough concentrations will be measured in order to determine volume of distribution

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ter Avest M, Langemeijer SMC, van den Heuvel LPWJ, Baas LM, van de Kar NCAJ, Ter Heine R. Model-Informed Precision Dosing of Eculizumab in Patients with Paroxysmal Nocturnal Hemoglobinuria. Clin Pharmacokinet. 2025 Aug;64(8):1139-1147. doi: 10.1007/s40262-025-01536-x. Epub 2025 Jun 25. PMID 40560515